CLINICAL TRIAL: NCT00949585
Title: Potassium Intake in Patients With Chronic Kidney Disease
Acronym: CKD-K
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Sharon Turban, Assistant Professor of Medicine, Division of Nephrology, Johns Hopkins University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AHA 0835162N
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: Chronic Kidney Disease; Hypertension
Keywords: randomized, controlled feeding study;; crossover design; potassium intake
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dietary potassium intake: 100 mmol/day (Other): Participants will be given one of two diets: one contains 100 mmol of potassium per day, and the other contains 40 mmol of potassium per day
  Interventions: Other: Dietary intake of potassium
- Dietary potassium intake: 40 mmol/day (Other): Diet containing 40 mmol/day of potassium
  Interventions: Other: Dietary intake of potassium

INTERVENTIONS:
Other: Dietary intake of potassium — Comparison of two diets: one contains 100 mmol potassium per day, and the other contains 40 mmol potassium per day

SUMMARY:
Chronic kidney disease is associated with high blood pressure, heart disease, and strokes. Potassium lowers blood pressure and may help prevent heart disease and strokes in the general population, but has not been well-studied in people with kidney disease. This study will look at the benefits and safety of two levels of potassium intake in patients with kidney disease. We expect that a higher level of potassium intake safely lowers blood pressure compared to a lower level of potassium intake. We hope that this and other research projects will help us to learn more so that guidelines can be created for potassium intake in patients with chronic kidney disease

DETAILED DESCRIPTION:
In individuals without chronic kidney disease (CKD), potassium (K) lowers blood pressure (BP) and may help prevent cardiovascular disease (CVD) and stroke. In animal models, K prevented kidney injury and decreased kidney inflammation. CKD patients may especially benefit from higher K intake, due to their high prevalence of hypertension, CVD, and stroke, and the possibility that K may retard CKD progression. Despite these potential benefits, there is great uncertainty about the optimal K intake in CKD patients. K is often restricted in these patients due to concerns about elevating serum K. However, renal K excretion does not appear to be substantially impaired until the glomerular filtration rate (GFR) is severely decreased (< 10-20 mL/min/1.73 m2). In this randomized feeding study with a two-period crossover design, the benefits and safety of 4 weeks of 100 mmol versus 40 mmol K/day in 26 non-diabetic adults with stage 3 CKD (estimated GFR 30-59 mL/min/1.73 m2) will be evaluated. After a one-week run-in period, all participants will be randomized to receive either a diet containing either 40 mmol K/day or 100 mmol K/day (within the current K/DOQI recommendations for K intake for stage 3 CKD) during period 1 (they will receive the other during period 2). The primary outcome variable is 24-hour ambulatory systolic BP. Secondary outcomes are other measures of peripheral BP, central BP, inflammatory markers, and serum K. We hope that this study will lead to a larger trial with sufficient power to examine the effects of increased K intake on clinical outcomes such as CKD progression. The ultimate goal of this effort is to develop the scientific basis for guidelines on K intake in CKD.

ELIGIBILITY:
Inclusion Criteria:

* Stage 3 chronic kidney disease (estimated glomerular filtration rate 30-59 mL/min/1.73 m2 by the 4-variable Modification of Diet in Renal Disease (MDRD) Study Equation
* Systolic blood pressure 120-159 mm Hg and diastolic blood pressure < 100 mm Hg
* Willingness to follow strict dietary rules for 9 weeks and to come to the clinical research unit at least 3 weekdays per week for one meal during the two study periods

Exclusion Criteria:

* Baseline serum potassium of at least 5.5 mEq/L
* Baseline serum potassium of less than 3.5 mEq/L
* Insulin-requiring or uncontrolled (HbA1C > 9 g/dL) diabetes mellitus
* Use of potassium supplements
* Use of digoxin
* Chronic disease(s) that may interfere with trial participation
* Pregnancy or lactation
* > 14 alcoholic drinks/week
* Major food allergies or intolerances

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
24-hour ambulatory systolic blood pressure | At screening, and at the end (4th week) of each intervention period

SECONDARY OUTCOMES:
other measures of peripheral blood pressure (other types of ambulatory blood pressure measurements as well as clinic blood pressure) | Ambulatory BP: same as primary outcome. Clinic BP: at screening, run-in, and weekly during intervention
measures of central blood pressure (pulse wave velocity and augmentation index) | at screening and at the end (4th week) of each intervention period
Serum potassium | At screening, run-in, and at least 3 times during each intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Turban, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University Pro Health Clinical Research Facility, Baltimore, Maryland, United States